CLINICAL TRIAL: NCT02424110
Title: Bipolar Radiofrequency Ablation Plus Endocardial Ablation Using Argon Beam Coagulator for Atrial Fibrillation Treatment in Patients With Rheumatic Heart Disease
Brief Title: Bipolar Radiofrequency Ablation Plus Argon Beam Coagulator Ablation for Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Mingwen Li, Resident surgeon in the Department of Cardiovascular Surgery of Xinqiao Hospital, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xqxwk_07
Record Dates: First submitted 2015-04-08; First posted 2015-04-22 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
Keywords: bipolar radiofrequency ablation; argon beam coagulator
MeSH Terms: conditions — Atrial Fibrillation | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Argon beam coagulator ablation group (Experimental): In the bipolar left atrial radiofrequency ablation, when the linear ablation was performed through along the lower edge of interatrial groove incision up to the mitral annulus, there is a gap between the ends of the ablation line and the mitral annulus And in the bipolar right atrial radiofrequency ablation, when the linear ablation was performed along the lower edge of the coronary sinus ostium up to the inferoseptal commissure and through the vertical incision on anterior wall of the right atrium up to the tricuspid annulus. There also have gaps between ends of the ablation line and the tricuspid annulus. In the experimental group the investigators plan to use conventional bipolar radiofrequency ablation and use argon beam coagulator to ablate these gaps.
  Interventions: Procedure: argon beam coagulator ablation; Device: argon beam coagulator （American，Valleylab）
- Bipolar radiofrequency ablation group (Experimental): Only use conventional bipolar radiofrequency ablation and do not deal with these gaps.
  Interventions: Procedure: bipolar radiofrequency ablation; Device: bipolar radiofrequency (AtricuteTM)

INTERVENTIONS:
Procedure: argon beam coagulator ablation — The investigators plan to use argon beam coagulator ablation plus bipolar radiofrequency ablation in the argon beam coagulator ablation group.
  Arms: Argon beam coagulator ablation group
Procedure: bipolar radiofrequency ablation — The investigators only use bipolar radiofrequency ablation in the left and right atrial radiofrequency ablation.
  Arms: Bipolar radiofrequency ablation group
Device: argon beam coagulator （American，Valleylab） — Argon beam coagulator（American，Valleylab）will be used in the argon beam coagulator ablation group
  Arms: Argon beam coagulator ablation group
Device: bipolar radiofrequency (AtricuteTM) — The investigators plan to use bipolar radiofrequency(AtricuteTM) in the bipolar radiofrequency group
  Arms: Bipolar radiofrequency ablation group

SUMMARY:
The objective of the study is to make up the technique blind spots of the bipolar radiofrequency ablation in the surgical treatment of atrial fibrillation with rheumatic heart disease by using argon beam coagulator. And to improve the rates of cardioversion of atrial fibrillation after surgery, to decrease the long-term recurrence rate of atrial fibrillation and to compare the early term and long term outcomes of bipolar radiofrequency ablation and bipolar radiofrequency plus argon beam coagulator ablation.

DETAILED DESCRIPTION:
Atrial fibrillation(AF) is the most common sustained arrhythmia. It can cause reduced heart function and increase the risk of thromboembolism. About 60% of patients with rheumatic heart disease have persistent AF.AF surgery is an effective intervention for patients with all types of AF undergoing concomitant cardiac surgery. AF surgery can reduce the risks of heart of stroke and heart failure and promote longer survival. Bipolar radiofrequency ablation is one of the most effective ways. But in the investigators' early study we find that there are technique blind spots in the left atrial ablation and right atrial ablation. In the bipolar left atrial linear ablation performed along the lower edge of interatrial groove incision up to the mitral annulus, there is a gap between the ends of the ablation line to the mitral annulus. And if the investigators use bipolar radiofrequency pliers it may injure the lcx left circumflex artery and left ventricular. In the bipolar right atrial radiofrequency ablation, the linear ablation performed along the lower edge of the coronary sinus ostium up to the inferoseptal commissure and the linear performed through the vertical incision on anterior wall of the right atrium up to the tricuspid annulus, there is also a gap between the end of the end of the ablation line and the tricuspid annulus. These gaps are one of factors of the recurrence of AF.

Argon beam coagulator is one of the most common hemostasis tools in heart surgery. It can also cause coagulation necrosis of the myocardium and do not do harm to the nearly myocardium the same as bipolar radiofrequency ablation. In the investigators' early study the investigators use the coagulation de plasma argon to burn the endocardium. And in the investigators' 6 mouth follow up, the rate of cardioversion is 90%. In this study the investigators plan to use argon beam coagulator to ablate these gaps.

The objective of the study is to make up the technique blind spots of the bipolar radiofrequency ablation in the surgical treatment of atrial fibrillation with rheumatic heart disease by using argon beam coagulator. And to improve the rates of cardioversion of atrial fibrillation after surgery, to decrease the long-term recurrence rate of atrial fibrillation and to compare the early term and long term outcomes of bipolar radiofrequency ablation and bipolar radiofrequency plusargon beam coagulator ablation.

ELIGIBILITY:
Inclusion Criteria:

* The patients got atrial fibrillation with rheumatic heart disease need surgical radiofrequency ablation treatment

Exclusion Criteria:

* left atrial diameter>65mm，
* sick sinus syndrome，
* atrioventricular block，
* ventricular tachycardia，
* reoperation patients，
* implantation of permanent pacemaker，
* NYHA(New York Heart Association) class IV，
* Malignant tumor, or other serious diseases which life expectancy < 1 year，
* Heating temperature above 38 degrees or active infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
electrocardiogram：rates of cardioversion of atrial fibrillation | 3 years after surgery
  The investigators plan to check the electrocardiogram of all the 200 individuals involved in our study 3 years after surgery to ensure the rate of cardioversion of atrial fibrillation

SECONDARY OUTCOMES:
surgery time | during surgery
cardiopulmonary bypass time | during surgery
long-term recurrence rate of atrial fibrillation | 3 years
complication after surgery | 3 years
  Number of adverse events as an assessment of complications after surgery
radiofrequency ablation time | during surgery
hospital stays | 4 weeks
  participants will be followed for the duration of hospital stay，an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, Study Director — Department of Cardiovascular Surgery, Xinqiao Hospital, Third Military Medical University
Locations (1):
- Lin Chen, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] [1] Hong L, Lin C, Yinbing X, et al. Early Efficacy Analysis of Biatrial Ablation versus Left and Simplified Right Atrial Ablation for Atrial Fibrillation Treatment in Patients with Rheumatic Heart Disease. Heart Lung Circ. 2015 [2] Hussein AA, Wazni OM, Harb S, Joseph L, Chamsi-Pasha M, Bhargava M,et al. Radiofrequency Ablation of Atrial Fibrillation in Patients With Mechanical Mitral Valve Prostheses. J Am Coll Cardio 2011;58:596-602 [3] PasicM, Bergs P, Muller P, et al. Intraoperative radiofrequencymaze ablation for trail fibrillation: the berlin modification [J]. Ann Thorac Surg,2001,72(5):1484-1490 [4] WilliamsM R, GarridoM, OzMC, et al. Alternative energy source for surgical atrial ablation [J].J Card Surg,2004,19(3):201-206 [5] Nitta T. Surgery for trail fibrillation: a worldwide review [J]. Semin Thorac Cardiovasc Surg, 2007, 19(1):3-8